CLINICAL TRIAL: NCT00667394
Title: A Phase 2 Trial of Tandutinib in Combination With Bevacizumab for Patients With Recurrent High-Grade Gliomas
Brief Title: Tandutinib Plus Bevacizumab to Treat Recurrent Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Katherine E. Warren, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 080101; 08-C-0101
Record Dates: First submitted 2008-04-25; First posted 2008-04-28 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-10

CONDITIONS: Glioblastoma; Gliosarcoma; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Anaplastic Mixed Oligoastrocytoma
Keywords: Brain Tumor; Chemotherapy; Radiation; Anti-Angiogenesis; Glioblastoma; Glioma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Astrocytoma; Oligodendroglioma; Brain Neoplasms; Glioma | interventions — Bevacizumab; tandutinib; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tandutinib & Bevacizumab in GBM Patients (Experimental): GBM (glioblastoma multiforme) Tandutinib 500 mg by mouth daily dose twice a day. Bevacizumab 10 mg/kg dose intravenous repeated once every 2 weeks.
  Interventions: Biological: Bevacizumab; Drug: MLN-518 (Tandutinib); Procedure: Quality-of-life assessment
- Tandutinib & Bevacizumab in AG Patients (Experimental): AG (anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic mixed oligoastrocytoma, and malignant astrocytoma NOS (not otherwise specified)) Tandutinib 500 mg by mouth daily dose twice a day. Bevacizumab 10 mg/kg dose intravenous repeated once every 2 weeks.
  Interventions: Biological: Bevacizumab; Drug: MLN-518 (Tandutinib); Procedure: Quality-of-life assessment

INTERVENTIONS:
Biological: Bevacizumab — Bevacizumab 10 mg/kg dose intravenous repeated once every 2 weeks.
Drug: MLN-518 (Tandutinib) — Tandutinib 500 mg by mouth daily dose twice a day.
Procedure: Quality-of-life assessment — Forty-five one-sentence questionnaire to assess health related quality of life in patients with brain cancer.
  Other Names: HRQL (health related quality of life)

SUMMARY:
Background:

In order to survive, brain tumors must have a network of blood vessels to supply it with oxygen and nutrients. The tumors produce substances that enable new blood vessels to form.

Tandutinib and Bevacizumab are experimental drugs that may prevent new blood vessel formation and thereby slow or stop tumor growth in the brain.

Objectives:

To determine the safety and side effects of Tandutinib in combination with Bevacizumab in patients with brain tumors.

To evaluate the response of brain tumors to treatment with Tandutinib and Bevacizumab.

Eligibility:

Patients 18 years of age and older with a malignant brain tumor for whom standard treatments (surgery, radiation and chemotherapy) are no longer effective.

Design:

Patients receive treatment in 4-week cycles as follows: Tandutinib by mouth twice a day every day and intravenous (through a vein) infusions of Bevacizumab over 90 minutes (or less if well tolerated) every 2 weeks. Treatment may continue for up to 1 year, and possibly longer, as long as there are no signs of tumor growth or serious treatment side effects.

Patients are evaluated with magnetic resonance imaging (MRI), computed tomography (CT) and positron emission tomography (PET) scans before starting treatment and then periodically to determine the response to treatment.

Patients have physical and neurological examinations every 4 weeks and blood tests every 2 weeks. They complete quality of life questionnaires every 4 weeks.

DETAILED DESCRIPTION:
Background

Bevacizumab is a monoclonal antibody directed against vascular- endothelial growth factor (VEGF), the major angiogenesis factor involved in high-grade glioma-mediated angiogenesis. Preclinical studies in our laboratory and others have shown potent antiglioma activity in vivo and early clinical trials of bevacizumab in combination with irinotecan and alone (National Institutes of Health (NIH) study) have demonstrated significant anti-vascular permeability and anti-glioma effects in patients with recurrent gliomas.

Tandutinib (MLN518) along with bevacizumab represents an attempt to further capitalize on the concept of targeting the tumor vasculature. Tandutinib is a small molecule inhibitor of fms-like tyrosine kinase receptor-3 (FLT3), platelet derived growth factor receptor (PDGFR), and cKIT (type III receptor tyrosine kinases). It has demonstrated anti-leukemic activity in patients with relapsed and refractory acute myeloid leukemia (AML) whose blasts contain an activating internal tandem duplication mutation of FLT3. However, in this study tandutinib is being added to bevacizumab primarily for its activity against the PDGFR and cKIT. Hannahan and colleagues have demonstrated the additional anti-tumor activity that results in vivo with combined inhibition of the vascular endothelial growth factor receptor (VEGFR) and PDGFR. The activity of PDGFR inhibition is hypothesized to result from its effect on pericytes, the cells that surround and support endothelial cells. These cells have abundant expression of PDGFR and require platelet-derived growth factor (PDGF)-PDGFR interaction for their normal function.

Objectives

To establish data regarding the anti-tumor activity of the combination of bevacizumab and tandutinib in patients with recurrent high-grade gliomas, as determined by progression-free-survival.

Eligibility

Patients with histologically proven recurrent malignant glioma are eligible for this study.

Design

Patients will receive tandutinib as a single agent at a daily dose of 500 mg PO bid for the first 14 days of treatment. Radiology: Prior to the first dose of tandutinib patients will undergo an MRI-perfusion scan and an FDG-PET scan. An MRI-perfusion scan will then be repeated between days 12-14 of the first 14 days of tandutinib monotherapy. On day 15, treatment with bevacizumab will be added to the ongoing treatment with tandutinib. Bevacizumab will be given intravenously in a dose of 10 mg/kg, repeated once every 2 weeks. After completion of the first 4 weeks of combined tandutinib and bevacizumab therapy (6 weeks after initiating treatment with tandutinib) considered the first cycle of therapy) the MRI-perfusion and fludeoxyglucose 18F-positron emission tomography (FDG-PET) scans will be repeated before the next dose of bevacizumab is given. Patients who are clinically/neurologically stable, and who have radiographically stable or responding disease at the end of that first cycle and every cycle thereafter (every 4 weeks), will continue treatment with tandutinib and bevacizumab. Magnetic resonance imaging (MRI)-perfusion scans will be repeated after the completion of every 4 weeks of therapy. A total of 80 patients will be enrolled to this study (GBM (glioblastoma multiforme)=40, AG=40)

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with histologically proven intracranial malignant glioma will be eligible for this protocol.

Malignant glioma includes glioblastoma multiforme (GBM), gliosarcoma, anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed oligoastrocytoma (AMO), or malignant astrocytoma NOS (not otherwise specified).

* Patients must have evidence for tumor progression by magnetic resonance imaging (MRI) or computed tomography (CT) scan.

This scan should be performed within 14 days prior to registration and on a fixed dose of steroids for at least 5 days.

If the steroid dose is increased between the date of imaging and registration a new baseline MRI/CT is required.

The same type of scan, i.e. MRI or CT must be used throughout the period of protocol treatment for tumor measurement.

* Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply:
* They have recovered from the effects of surgery.
* Residual disease following resection of recurrent tumor is not mandated for eligibility into the study.

To best assess the extent of residual disease post-operatively, a CT/ MRI should be done:

* no later than 96 hours in the immediate post-operative period or
* at least 4 weeks post-operatively, and
* within 14 days of registration, and
* on a steroid dosage that has been stable for at least 5 days.

  * If the 96 hour scan is more than 21 days before registration, the scan needs to be repeated.

If the steroid dose is increased between the date of imaging and registration, a new baseline MRI/CT is required on a stable steroid dosage for at least 5 days.

* Patients must have progressed after radiation therapy and must have an interval of greater than or equal to 4 weeks from the completion of radiation therapy to study entry.
* All patients or their previously designated durable power of attorney (DPA) (if the patient is deemed by the treating physician to be impaired or questionably impaired in such a way that the ability of the patient to give informed consent is questionable) must sign an informed consent indicating that they are aware of the investigational nature of this study.
* Patients must be greater than or equal to 18 years old, and with a life expectancy greater than 8 weeks.
* Patients must have a Karnofsky performance status of greater than or equal to 60.
* Patients must have recovered from the toxic effects of prior therapy: 2 weeks from any investigational agent, 4 weeks from prior cytotoxic therapy, two weeks from vincristine, 6 weeks from nitrosoureas, 3 weeks from procarbazine administration, and 1 week for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count). Any questions related to the definition of non-cytotoxic agents should be directed to the Study Chair.
* Patients must have adequate bone marrow function (white blood cell (WBC) greater than or equal to 3,000/microl, Absolute neutrophil count (ANC) greater than or equal to 1,500/mm^3, platelet count of greater than or equal to 100,000/mm^3, and hemoglobin greater than or equal to 10 gm/dl), adequate liver function (serum glutamic oxaloacetic transaminase (SGOT) and bilirubin less than 2 times upper limit of normal (ULN)), and adequate renal function (creatinine less than 1.5 mg/dL and/or creatinine clearance greater than or equal to 60 cc/min) before starting therapy.

Serum sodium, calcium, potassium, chloride, and magnesium must be in normal limits.

These tests must be performed within 14 days prior to registration. Eligibility level for hemoglobin may be reached by transfusion.

* Patients must not have any significant medical illnesses that, in the investigator's opinion, cannot be adequately controlled with appropriate therapy or would compromise the patients' ability to tolerate this therapy
* This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender. No exclusion to this study will be based on race. Minorities will actively be recruited to participate.
* Creatinine clearance or calculated creatinine clearance greater than or equal to 60 mL/minute.
* Patients must practice adequate contraception.
* Head CT Scan without contrast (to rule out significant acute hemorrhage) within 7 days prior to starting treatment.
* A 12 lead electrocardiogram (ECG) to be performed within 2 weeks of trial entry with corrected QT interval (QTc) less than 460 msec.

EXCLUSION CRITERIA:

* Patients who, in the view of the treating physician, have significant active cardiac, hepatic, renal, or psychiatric diseases are ineligible.
* No concurrent use of other standard chemotherapeutics or investigative agents.
* Patients known to have a malignancy that has required treatment in the last 12 months and/or is expected to require treatment in the next 12 months (except non-melanoma skin cancer or carcinoma in-situ in the cervix).
* Patients who have an active infection.
* Pregnant (positive pregnancy test) or nursing women. Fertile men and women must agree to use adequate contraceptive measures during study therapy and for at least 6 months after the completion of tandutinib plus bevacizumab therapy.
* Patients who have any disease that will obscure toxicity (i.e. vasculitis, congenital hypercoaguability syndromes, uncontrolled primary hypertension, idiopathic thrombocytopenia).
* Evidence of significant recent hemorrhage on mandatory CT scan (defined as 1 cm or more of acute blood) of the brain within 7 days of patient accrual with the following exceptions: resolving hemorrhagic changes related to surgery, and/or presence of punctate hemorrhages in the tumor.
* Concurrent anti-coagulation or anti-platelet medication (including aspirin, non-steroidal anti-inflammatories, cyclooxygenase -2 (COX-2) inhibitors).
* Serious or non-healing wound, ulcer or bone fracture.
* Proteinuria at screening as demonstrated by either:
* Urine protein:creatinine (UPC) ratio greater than or equal to 1.0 at screening OR
* Urine dipstick for proteinuria greater than or equal to 2+ (patients discovered to have greater than or equal to 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate less than or equal to 1g of protein in 24 hours to be eligible).
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months
* Invasive procedures defined as follows:
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to Day 1 therapy
* Anticipation of need for major surgical procedures during the course of the study
* Core biopsy within 7 days prior to D1 therapy
* Patients with clinically significant cardiovascular disease
* History of cerebrovascular accident (CVA) or transient ischemic attack within 6 months
* Inadequately controlled hypertension (defined as systolic blood pressure greater than 160 and/or diastolic blood pressure greater than 100 mmHg on antihypertensive medications)
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* Myocardial infarction or unstable angina within 6 months
* New York Heart Association Grade II or greater congestive heart failure
* Serious cardiac arrhythmia requiring medication
* Unstable angina pectoris
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Prothrombin time (PT)/partial thromboplastin time (PTT) greater than1.5 time the upper limit of normal
* Patients with known hypersensitivity of Chinese hamster ovary cell products or other recombinant human antibodies
* Inability to take oral medication
* Known gastrointestinal disease or history of gastrointestinal surgery that could interfere with the absorption of orally administered medication.
* Ongoing vomiting
* Active cardiac disease as defined by:
* Significant cardiac event (including symptomatic heart failure or evidence of cardiac ischemia within 3 months of first dose or presence of any cardiac disease that in the opinion of the Investigator increases the risk of ventricular arrhythmia.
* Clinically significant arrhythmia (multifocal premature ventricular contraction [PVC], bigeminy, trigeminy, ventricular tachycardia, bradycardia) that is symptomatic or requires treatment (Common Terminology Criteria for Adverse Events (CTCAE) grade 3), or asymptomatic sustained ventricular tachycardia.
* Previous history of QTc prolongation with other medication.
* Congenital long QT syndrome
* QTc with Bazett's correction that is unmeasurable, or greater than or equal to 460 msec on screening ECG. If a patient has QTc greater than or equal to 460 msec on screening ECG, a second screen ECG may be repeated at least 24 hours apart. The average QTc from the 2 screening ECGs must be less than 460 msec in order for the patient to be eligible for the study. If the patient meets eligibility requirements in this way, the 'baseline' QTc for this patient will be the average of the 3 ECGs (screen 1, screen 2, and pre- 1 first dose).
* Previous history of left ventricular ejection fraction (LVEF) less than 45 percent as measured by multi-gated acquisition scan (MUGA) or by echocardiogram (ECHO) for patients with previous anthracycline therapy (total dose greater than 450 mg/m^2 or significant cardiovascular disease or chest irradiation, as determined by the investigator.
* A cardiac arrhythmia serious enough to require therapy (i.e. drugs, acquired immune deficiency (AID)), angina, symptomatic congestive heart failure and/or a cardiac ejection fraction less than 45 percent.
* Prior serious cardiac disease defined as prior coronary bypass surgery, angioplasty, or prior myocardial infarction unless a recent cardiac evaluation (within the last 3 months) demonstrated no significant coronary artery disease (i.e. a negative stress test) and no myocardial wall dysfunction.
* Concurrent use of other standard chemotherapeutics or investigative agents or vasoconstrictors for the treatment of migraine (ergotamine, zolmitriptan, sumatriptan) because of the potential for exacerbation of coronary vasoconstriction.
* Known or suspected primary muscular or neuromuscular disease (e.g. muscular dystrophy, myasthenia gravis). This does not include steroid myopathy.
* Prior treatment with bevacizumab is not permitted.
* Concurrent use of other drugs that have been shown to potentially prolong the QTc interval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Fine, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bigner SH, Bjerkvig R, Laerum OD. DNA content and chromosomal composition of malignant human gliomas. Neurol Clin. 1985 Nov;3(4):769-84. PMID 3001489
- [Background] Moss AR. Occupational exposure and brain tumors. J Toxicol Environ Health. 1985;16(5):703-11. doi: 10.1080/15287398509530780. PMID 4093991
- [Background] Bovet P, Lob M. [Cancer mortality among the workers of a Swiss rubber goods factory. Epidemiological study, 1955-75]. Schweiz Med Wochenschr. 1980 Aug 30;110(35):1277-87. French. PMID 6999620
- [Derived] Odia Y, Sul J, Shih JH, Kreisl TN, Butman JA, Iwamoto FM, Fine HA. A Phase II trial of tandutinib (MLN 518) in combination with bevacizumab for patients with recurrent glioblastoma. CNS Oncol. 2016;5(2):59-67. doi: 10.2217/cns-2015-0010. Epub 2016 Feb 10. PMID 26860632
- [Derived] Odia Y, Shih JH, Kreisl TN, Fine HA. Bevacizumab-related toxicities in the National Cancer Institute malignant glioma trial cohort. J Neurooncol. 2014 Nov;120(2):431-40. doi: 10.1007/s11060-014-1571-6. Epub 2014 Aug 7. PMID 25098701
- [Derived] Lehky TJ, Iwamoto FM, Kreisl TN, Floeter MK, Fine HA. Neuromuscular junction toxicity with tandutinib induces a myasthenic-like syndrome. Neurology. 2011 Jan 18;76(3):236-41. doi: 10.1212/WNL.0b013e3182074a69. PMID 21242491
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-C-0101.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Tandutinib & Bevacizumab in AG Patients: AG (anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic mixed oligoastrocytoma, and malignant astrocytoma NOS (not otherwise specified )) Tandutinib 500 mg by mouth daily dose twice a day. Bevacizumab 10 mg/kg dose intravenous repeated once every 2 weeks
Period: Overall Study
Arm/Group | Tandutinib & Bevacizumab in GBM Patients | Tandutinib & Bevacizumab in AG Patients
Started | 41 | 1
Completed | 37 | 1
Not Completed | 4 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Progressive disease | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tandutinib & Bevacizumab in GBM Patients | Tandutinib & Bevacizumab in AG Patients | Total
Number analyzed (Participants) | 41 | 1 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 1 | 37
  >=65 years | 5 | 0 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.16 (11.52) | 63 (0) | 54.37 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 0 | 12
  Male | 29 | 1 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 38 | 1 | 39
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 0 | 3
  White | 32 | 1 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 41 | 1 | 42

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 6 Months
Description: Percentage of participants with progression free survival at 6 months. Progression is defined as a 25% increase in the sum of all measurable lesions (or two largest lesions if too numerous) over the smallest sum observed (over baseline if no decrease), clear worsening of any evaluable disease, appearance of any new lesion/site, or failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: 6 months
Measure: Median (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Tandutinib & Bevacizumab in GBM Patients | Tandutinib & Bevacizumab in AG Patients
Number analyzed (Participants) | 37 | 0
Percentage of participants | 23 [12 to 37] |

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 45 months
Measure: Number; unit: Participants
Arm/Group | Tandutinib & Bevacizumab in GBM Patients | Tandutinib & Bevacizumab in AG Patients
Number analyzed (Participants) | 41 | 1
Participants | 40 | 1

ADVERSE EVENTS:
Arm/Group | Tandutinib & Bevacizumab in GBM Patients | Tandutinib & Bevacizumab in AG Patients
Serious Adverse Events (participants affected / at risk) | 15/41 | 0/1
Other Adverse Events (participants affected / at risk) | 41/41 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tandutinib & Bevacizumab in GBM Patients (N=41) | Tandutinib & Bevacizumab in AG Patients (N=1)
Death not associated with CTCAE term: Death Progression NOS (General disorders) | 1 (1) | 0 (0)
Dermatology/Skin - Other (Specify, keratosis & dermal hematoma) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hemorrhage, CNS (Nervous system disorders) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Abdomen NOS (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Colon (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Lung (pneumonia) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Pleura (empyema) (Infections and infestations) | 1 (1) | 0 (0)
Infection with unknown ANC::Lung (pneumonia) (Infections and infestations) | 1 (1) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy)::Extremity-lower (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain-Other (Specify, lower extremities) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy)::Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain::Head/headache (Nervous system disorders) | 1 (1) | 0 (0)
Perforation, GI::Stomach (Gastrointestinal disorders) | 1 (1) | 0 (0)
Platelets (Investigations) | 1 (1) | 0 (0)
Prolonged QTc interval (Investigations) | 1 (1) | 0 (0)
Psychosis (hallucinations/delusions) (Psychiatric disorders) | 1 (1) | 0 (0)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 5 (7) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 0 (0)
Perforation, GI::Colon (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tandutinib & Bevacizumab in GBM Patients (N=41) | Tandutinib & Bevacizumab in AG Patients (N=1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 4 (6) | 0 (0)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 16 (26) | 0 (0)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Alkaline phosphatase (Investigations) | 6 (7) | 0 (0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Bilirubin (hyperbilirubinemia) (Investigations) | 4 (6) | 0 (0)
Blood/Bone marrow - Other (Specify, elevated eosinophils) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Creatinine (Investigations) | 2 (4) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dermatology/Skin - Other (Specify,hyperpigmentation 1; laceration) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 31 (40) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Edema::head and neck (General disorders) | 17 (21) | 0 (0)
Edema: limb (General disorders) | 9 (9) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 21 (30) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glucose, serum-low (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hemoglobin (Investigations) | 14 (22) | 1 (2)
Hemoglobinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemorrhage, GI::Anus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhage, GI::Rectum (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hemorrhage, pulmonary/upper respiratory::Nose (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hemorrhage/Bleeding - Other (hemorrhage into sclera) (Eye disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 16 (24) | 1 (1)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Infection with unknown ANC::Lip/perioral (Infections and infestations) | 1 (1) | 0 (0)
Keratitis (corneal inflammatory/corneal ulceration) (Eye disorders) | 1 (1) | 0 (0)
Leukocytes (total WBC) (Investigations) | 21 (69) | 0 (0)
Lymphedema-related fibrosis (Vascular disorders) | 1 (1) | 0 (0)
Lymphopenia (Investigations) | 23 (73) | 0 (0)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy)::Extraocular (Eye disorders) | 1 (1) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy)::Extremity-lower (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy)::Whole body/generalized (Musculoskeletal and connective tissue disorders) | 7 (12) | 0 (0)
Nail changes (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 22 (27) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 13 (49) | 0 (0)
Pain::Other (Specify, left arm (phlebotomy pain)) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain::Chest wall (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain::Head/headache (Nervous system disorders) | 6 (7) | 0 (0)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain::Neck (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain::Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 15 (35) | 1 (3)
Platelets (Investigations) | 17 (31) | 0 (0)
Prolonged QTc interval (Investigations) | 21 (51) | 0 (0)
Proteinuria (Renal and urinary disorders) | 18 (21) | 1 (2)
Pyramidal tract dysfunction (e.g., increased tone, hyperflexia, positive Babinski, decreased fine mo (Nervous system disorders) | 1 (1) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Sodium, serum-low (hypernatremia) (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (4) | 0 (0)
Vision-blurred vision (Eye disorders) | 4 (4) | 0 (0)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (6) | 0 (0)
Weight gain (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No